CLINICAL TRIAL: NCT02051478
Title: CHANGES IN PRESSURE PAIN SENSITIVITY AND NECK PAIN AFTER THORACIC THRUST MANIPULATION OR NON-THRUST MOBILIZATION IN PATIENTS WITH MECHANICAL NECK PAIN
Brief Title: Thoracic Manipulation and Mobilization for Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, César Fernández-de-las-Peñas, Head Division, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: URJC2012/11
Record Dates: First submitted 2014-01-28; First posted 2014-01-31 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Neck Pain
Keywords: manipulation; mobilization; spine; pressure pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thoracic manipulation (Experimental): A high-velocity, end range, anterior-posterior thrust applied through the elbows to the mid-thoracic spine will be applied.
  Interventions: Other: Thoracic manipulation
- Thoracic mobilization (Active Comparator): Patients will receive 20 seconds bouts of grade III-IV of central posterior-anterior (PA) non-thrust mobilization from T3 to T6 spinous process as described by Maitland et al for an overall intervention time of approximately 2 minutes
  Interventions: Other: Thoracic mobilization

INTERVENTIONS:
Other: Thoracic mobilization — Patients will receive 20 seconds bouts of grade III-IV of central posterior-anterior (PA) non-thrust mobilization from T3 to T6 spinous process as described by Maitland et al for an overall intervention time of approximately 2 minutes
  Arms: Thoracic mobilization
Other: Thoracic manipulation — A high-velocity, end range, anterior-posterior thrust applied through the elbows to the mid-thoracic spine will be applied
  Arms: Thoracic manipulation

SUMMARY:
The purpose of this randomized clinical trial was to examine the widespread effects of thoracic spine thrust manipulation and thoracic non-thrust mobilization on pressure pain sensitivity and neck pain intensity in patients with chronic mechanical neck pain.

ELIGIBILITY:
Inclusion Criteria:

* mechanical idiopathic neck pain
* bilateral pain symptoms
* chronic pain (>3 months of duration)

Exclusion Criteria:

* whiplash injury
* previous spine surgery
* diagnosis of cervical radiculopathy or myelopathy
* diagnosis of fibromyalgia
* having undergone any physical therapy intervention in the previous year
* pregnancy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in Pressure pain thresholds | Change between baseline and 1o minutes immediate after the intervention
  The amount of pressure applied for the pressure sensation to first change to pain will be assessed with an electronic algometer (Somedic AB, Farsta, Sweden) over the C5-C6 zygapophyseal joint, second metacarpal and tibialis anterior muscle

SECONDARY OUTCOMES:
Change in Neck pain intensity | Change between baseline and 1o minutes immediate after the intervention
  Participants will rate the intensity of their neck pain at rest on an 11-point numerical pain rate scale (NPRS, 0: no pain, 10: maximum pain)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Salom.Moreno, PT, PhD, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain